CLINICAL TRIAL: NCT02142231
Title: Acupuncture Randomized Trial for Preventing Test Anxiety
Brief Title: AcuTA: Acupuncture in Test Anxiety
Acronym: AcuTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Goethe University (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Dr. Johannes Fleckenstein, Dr. med., Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AcuTA
Record Dates: First submitted 2014-04-24; First posted 2014-05-20 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2015-01

CONDITIONS: Test Anxiety; Experimental Setting (Trier Social Stress Test TSST)
Keywords: acupuncture; test anxiety; neuroenhancer; placebo
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laser Acupuncture (Placebo Comparator): Subjects and Therapists are blinded. Instead of a real Laser Acupuncture device (able to elicit physiologic responses) them is given a sham-laser device only radiating non-energetic red LED-light. Without palpation, therapists treat the acupoint Heart 7, on both wrists, each for 1 minute, with additional 18 minutes of resting time after.
  Interventions: Device: Laser Acupuncture
- Acupuncture (Active Comparator): Acupuncture at the acupoint Heart 7, on both wrists, each for 1 minute, eliciting a deqi-response, additional stimulation and total needle-in time of 20 minutes (2 minutes treatment and 18 minutes of resting time)
  Interventions: Device: Acupuncture

INTERVENTIONS:
Device: Acupuncture — Sterile Acupuncture Needles (Seirin (R) 0.15x0.2) will be used, Needles are inserted for approx. 0.5-1 cm until deqi response is elicited
  Arms: Acupuncture
Device: Laser Acupuncture — Therefore a laser irradiation is faked, approaching a nonfunctioning laser pen, which has been deactivated by the manufacturer (3B Scientific GmbH, Hamburg, Germany). Only red light is emitted. To further emphasize the imaginary power of this sham procedure, visual and acoustic signals accompany the red light emission. Patients are treated at the same acupuncture points as in the acupuncture group for one minute without skin contact. The resting time after treatment is 18 minutes.
  Arms: Laser Acupuncture

SUMMARY:
Test anxiety is a well-known phenomenon in general population, but only few scientific advances have been made in order to fully understand and prevent this circumstance.

The number of students which use neuro enhancement to improve their performance and to prevent test anxiety, is increasing. A US-survey estimated that almost 7% of students in US universities have used prescription stimulants against anxiety, and that on some campuses, up to 25% of students had used them in the past year.

Acupuncture might act as an alternate. Several trials could demonstrate, that different forms of acupuncture could relieve symptoms of pre-exam anxiety syndrome significantly and that this therapy was highly safe. In special, the investigation of single point effects in test anxiety could be of general interest. The acupuncture point with the most convincing evidence up to date is Heart 7. Yet, its effectiveness has mainly been chosen in combination with other acupuncture points and not as single remedy in test anxiety. Therefore we establish a trial investigating the immediate needling effects at Heart 7 on the reduction of test anxiety.

Therefore qe implemented a validated stress test, the Trier Social Stress Test TSST, which is known to provoke serious stress responses in healthy subjects. 24 medical students with test anxiety in there history will be randomised to two interventional groups (verum acupuncture and laser acupuncture), being treated and then pass this test. Main outcome is the increase of cortisol in saliva, which is the standardized measure of stress response used in this paradigm.

ELIGIBILITY:
Inclusion Criteria:

* Test Anxiety in the clinical history
* Male medical students 3rd to 5th year
* Compliance
* Age > 18 years
* Smoking cessation for 24 hours

Exclusion Criteria:

* Severe physical or psychical illness
* Psychiatric record in medical history
* Continuous uptake of antipsychiatric medication, tranquilizers or neuro-enhancers
* Acupuncture treatment within the last 4 weeks
* Hang-over
* Drug consumption
* Smoking (> 5 cigarettes/ day)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Cortisol in saliva | 8 timepoints (in minutes: -40;-10;+10;+20;+30;+40;+55;+70)
  Saliva samples will be obtained at above mentioned intervals for subsequent analysis of cortisol a in saliva. The stress model used in this trial is supposed to elevate cortisol in saliva 3-5 fold in controls.

SECONDARY OUTCOMES:
Test Anxiety on a Visual Analogue Scale | 4 timepoints (in minutes: -40;-10;+20;+55)
  Visual Analogue Scale (ranging 0 to 10, with 10 being most anxious)
Primary Appraisal Secondary Appraisal | 2 timepoints (-40 and +10 minutes)
  validated questionnaire
Multidimensional Mood State Questionnaire | 4 timepoints )in minutes: -40;-10;+10;+20)
  validated questionnaire
State Trait Anxiety Questionnaire | 3 timepoints (in minutes: -40;-10;+10)
  validated questionnaire
alpha amylase in saliva | 6 timepoints (in minutes: -40;-10;+10;+20;+30;+55)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical School, University of Regensburg, Germany, Bavaria, Germany